CLINICAL TRIAL: NCT00864253
Title: An Open-Label, Multicenter, Phase III Trial of ABI-007 vs Dacarbazine in Previously Untreated Patients With Metastatic Malignant Melanoma
Brief Title: A Trial of ABI-007 Versus Dacarbazine in Previously Untreated Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA033
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Malignant; Abraxane; ABI-007; Dacarbazine; Dtic-Dome
MeSH Terms: conditions — Melanoma | interventions — Albumin-Bound Paclitaxel; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABI-007 (Experimental): Treatment Arm A (ABI-007): Patients who receive ABI-007 will be dosed intravenously over approximately 30 minutes without steroid pre-medication and without G-CSF prophylaxis (unless modified as described below). ABI-007 150 mg/m2 will be administered on Days 1, 8, and 15 every 4 weeks.
  Interventions: Drug: ABI-007
- Dacarbazine (Active Comparator): Treatment Arm B (dacarbazine): Patients who receive dacarbazine will be dosed intravenously at 1000 mg/m2 on Day 1 with steroid and antiemetic pre-medication. Treatment will be repeated every 21 days.
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: ABI-007 — Patients who receive ABI-007 will be dosed intravenously over approximately 30 minutes without steroid pre-medication and without G-CSF prophylaxis (unless modified as described below). ABI-007 150 mg/m2 will be administered on Days 1, 8, and 15 every 4 weeks.
  Other Names: Abraxane
  Arms: ABI-007
Drug: Dacarbazine — Patients who receive dacarbazine will be dosed intravenously at 1000 mg/m2 on Day 1 with steroid and antiemetic pre-medication. Treatment will be repeated every 21 days.
  Other Names: Dtic-Dome, DTIC-Dome
  Arms: Dacarbazine

SUMMARY:
The main purpose of this research study is to compare the safety, tolerability, and anti tumor activity of an investigational drug, ABI-007 versus Dacarbazine in patients with metastatic melanoma who have not previously received chemotherapy. ABI-007 is a new preparation of the active drug paclitaxel. It contains the same medication as the prescription chemotherapy drug Abraxane®. Abraxane® is approved by the FDA for the treatment of metastatic breast cancer after failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy. Dacarbazine is approved by the FDA for the treatment of melanoma. In this study, ABI-007 and Dacarbazine will be tested as therapy for people who have not yet had any cancer treatment for the diagnosis of metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cutaneous malignant melanoma with evidence of metastasis (Stage IV).
* No prior cytotoxic chemotherapy for metastatic malignant melanoma is permitted. Prior treatment with kinase inhibitors or cytokines is permitted.
* No prior adjuvant cytotoxic chemotherapy is permitted. Prior adjuvant therapy with interferon, Granulocyte-macrophage colony-stimulating factor (GM-CSF) and/or vaccines is permitted.
* Male or non-pregnant and non-lactating female, and ≥ 18 years of age. If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test Beta human chorionic gonadotropin (ß-hCG) within 72 hours prior to first study drug administration. If sexually active, the patient must agree to utilize contraception considered adequate and appropriate by the investigator.
* No other current active malignancy within the past 3 years.
* Radiographically-documented measurable disease (defined by the presence of at least 1 radiographically documented measurable lesion
* Patient has the following blood counts at Baseline:
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9 cells/L;
* platelets ≥ 100 x 10^9 cells/L;
* Hemoglobin (Hgb) ≥ 9 g/dL.
* Patient has the following blood chemistry levels at Baseline:
* Aspartate aminotransferase(AST) glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≤ 2.5x upper limit of normal range (ULN); ≤ 5.0 xULN if hepatic metastases present;
* total bilirubin ≤ ULN;
* creatinine ≤ 1.5 mg/dL.
* Lactate Dehydrogenase (LDH) ≤ 2.0 x ULNa
* Expected survival of > 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria:

* History of or current evidence of brain metastases, including leptomeningeal involvement.
* Patient has pre-existing peripheral neuropathy of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Scale of Grade ≥ 2.
* Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.
* Patient has a clinically significant concurrent illness.
* Patient is, in the investigator's opinion, unlikely to be able to complete the study through the End of Study (EOS) visit.
* Patient is currently enrolled, or will enroll in a different clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study. Marker studies or studies evaluating biological correlates are permitted.
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2014-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Hersh, MD, Principal Investigator — University of Arizona; Ileana Elias, MD, Study Director — Celgene Corporation
Locations (112):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AZ Cancer Ctr, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Genesis Cancer Ctr - Hot Springs, Hot Springs, Arkansas
  - University of Arkansa for Medical Sciences, Little Rock, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - San Diego Pacific Oncology and Hematology Associates, Encinitas, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - University of CA Los Angeles, Los Angeles, California
  - St. Mary's Medical Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Baptist Cancer Institute, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Miami Hospital and Clincs/SCCC, Miami, Florida
  - Waren Billhartz Cancer Center, Maryville, Illinois
  - Indiana University, Indianapolis, Indiana
  - IA Blood and Cancer Care, PLC, Cedar Rapids, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. John's Medical Research, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Atlantic Melanoma Center, Morristown, New Jersey
  - Piedmont Hematology, Winston-Salem, North Carolina
  - OH State University Arthur G. James Cancer Hospital, Columbus, Ohio
  - Integris Cancer Institute of OK, Oklahoma City, Oklahoma
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Mary Crowley Research Center, Dallas, Texas
  - Univ of TX MD Anderson Cancer Ctr, Houston, Texas
  - Univ of TX Med School at Houston, Houston, Texas
  - Covenant Health System DBA Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Hope Oncology, Richardson, Texas
  - Utah Cancer Specialist, Salt Lake City, Utah
  - Univ. of Washington Medical Center/Seattle Cancer Care Alliance, Seattle, Washington
  - Evergreen Hematology & Oncology, Spokane, Washington
- Australia (8):
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Sydney West Cancer Trials Centre/Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Department of Medical Oncology, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA, Centre for the Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency-Fraser Valley Ctr., Surrey, British Columbia
  - BC Cancer Agency-Vancouver, Vancouver, British Columbia
  - BC Cancer Agency-Vancouver Island Ctr., Victoria, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Missiauga, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Dept. of Oncology Clinical Research Program, Montreal, Quebec
- France (13):
  - Hopital Saint Andre' CHU de Bordeaux, Bordeaux
  - Centre Hospitaller Universitaire de Grenoble, Grenoble
  - CHRU Hopital Claude Huriez, Lile Cedax
  - Hopital Dypuytren-CHU de Limoges, Limoges
  - Centre Leon Berad, Lyon
  - Hopital Sainte Marguerite, Marseille
  - CHU Hopital Saint Eloi, Montepellier Cedex 5
  - Centre Regional Val d' Aurelle Paul Lamarque, Montpellier
  - Hopital de 1 Archet 2, Nice
  - Hopital Bichat, Paris
  - Groupe hospitalier Cochin-St. Vincent de Paul, Paris
  - Hopital Saint-Louis, Paris
  - Institut Gustave Roussy (IGR) Centre de Lutte Contre le Canc, Villejuif
- Germany (16):
  - Universitaetsklinkum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinkum Heidelberg, Heidelber, Baden-Wurttemberg
  - Universitaetsklinkum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinkum Wuerzburg PS, Würzburg, Bavaria
  - Universitaetsklinkum Hamburg-Eppendorf, Hamburg, Hamburg
  - Univeritaetsklinkum Goettingen, Gottington, Lower Saxony
  - Medizinische Hochschuke Hannover, Hanover, Lower Saxony
  - St. Josef-Hospital, Bochum, Northwest
  - Universitaetklinkum Koeln, Cologne, Northwest
  - Universitaetsklinkum Essen, Essen, Northwest
  - Universitaetsklinkum Dresden, Dresden, Saxony
  - Universitaetsklinkum Schegwig-Holstein, Keil, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin, Berlin, State of Berlin
  - UniversitawtsklinKum Jena, Jena, Strasse 35
  - Universitaesklinkum Leipzig, Leipzig
  - Universitaetsklinkum Mainz, Mainz
- Italy (9):
  - Istituto Tumori "Giovanni Paolo II", Bari, BA
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei T, Meldola, FC
  - IST-Istituto Nazionale per la Ricera sul Cancro, Genova, GE
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Nazionale Tumori, Milan, MI
  - IOV-Instituto Oncologico IRCCS, Padua, PD
  - Azienda Ospedaliera Universitaria Sense, Siena, SI
  - Ist. Naz. per lo studio e la cura dei tumori G. Pascale, Napoli
  - Ospedale S. Chiara, Pisa
- Netherlands (3):
  - Medisch Centrum Alkmaar, Alkmaar
  - Rijnstate ziekenhuis Arnhem, Amhem
  - Erasmus MC ae" Daniel den Hoed, Rotterdam
- Spain (4):
  - H Clinic i Provincial, Barcelona
  - H CLINIC I Provincial, Barcelona
  - H Clinico San Carlos, Madrid
  - Corporacion Sanitaria Parc Tauli, Sabadell
- United Kingdom (9):
  - Broomfield Hospital, Chelmsford, Essex
  - Velindre Hospital, Cardiff, GLAM
  - St. George's Hospital, London, GT Lon
  - Nottingham University Hospitals NHS Trust, Nottingham, NOTT
  - Singleton Hospital, Sothwest Wales Inst., Swansea, S GLAM
  - Univ Hospital of North Staffordshire, Stroke on Kent, Staffs
  - Weston Park Hospital, Sheffield, Syorks
  - Newcross Hospital, Wolverhampton, Wstmid
  - Royal Marsden Hospital London, London

REFERENCES:
- [Background] Hersh EM, Del Vecchio M, Brown MP, Kefford R, Loquai C, Testori A, Bhatia S, Gutzmer R, Conry R, Haydon A, Robert C, Ernst S, Homsi J, Grob JJ, Kendra K, Agarwala SS, Li M, Clawson A, Brachmann C, Karnoub M, Elias I, Renschler MF, Hauschild A. A randomized, controlled phase III trial of nab-Paclitaxel versus dacarbazine in chemotherapy-naive patients with metastatic melanoma. Ann Oncol. 2015 Nov;26(11):2267-74. doi: 10.1093/annonc/mdv324. Epub 2015 Sep 26. PMID 26410620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted by investigators in 9 countries: Australia, Canada, France, Germany, Italy, Netherlands, Spain, United Kingdom and the United States (US) and treatment was given on an outpatient basis. First participant enrolled 30 April 2011, last participant enrolled June 2011..
Pre-assignment Details: Participants were randomized in a 1:1 ratio. Randomization was stratified based on metastatic stage (M1a, M1b, and M1c), region (North America, Western Europe and Australia), and baseline lactate dehydrogenase (LDH) (< 0.8 * ULN, 0.8-1.1 * ULN, >1.1-2 * ULN).
Groups:
- ABI-007 150mg/m^2: ABI-007 150mg/m^2 intravenously over approximately 30 minutes on Days 1, 8 and 15 of each 28 day cycle
- Dacarbazine 1000mg/m^2: Dacarbazine 1000mg/m^2 intravenously over approximately 30-60 minutes on Day 1 of each 21 day cycle.
Period: Overall Study
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Started | 264 | 265
Treated | 257 | 258
Completed | 165 (Completed = defined as discontinuation due to progressive disease) | 207 (Completed = defined as discontinuation due to progressive disease)
Not Completed | 99 | 58
Not completed — Adverse Event | 56 | 11
Not completed — Unrelated Adverse Event | 3 | 1
Not completed — Physician Decision | 11 | 15
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 18 | 18
Not completed — Death | 1 | 0
Not completed — Ongoing | 2 | 3
Not completed — Untreated | 7 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population consisted of all randomized participants regardless of whether the participant received any study drug or had any efficacy assessments collected.
Groups:
- Dacarbazine Arm B 1000mg/m^2: Dacarbazine 1000mg/m^2 intravenously over approximately 30-60 minutes on Day 1 of each 21 day cycle.
- Total: Total of all reporting groups
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine Arm B 1000mg/m^2 | Total
Number analyzed (Participants) | 264 | 265 | 529
Age, Continuous [Median (Full Range); unit: years] | 62.0 (13.44) [21 to 85] | 64.0 (12.06) [28 to 87] | 63.0 (12.85) [21 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 91 | 182
  Male | 173 | 174 | 347
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — ECOG-Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = Fully Active | 195 | 181 | 376
    1= Restrictive but Ambulatory | 68 | 82 | 150
    2 = Ambulatory but Unable to Work | 1 | 2 | 3
    3 = Limited Self-Care | 0 | 0 | 0
    4 = Completely Disabled | 0 | 0 | 0
Baseline Lactate Dehydrogenase value [Number; unit: participants] — The serum level of Lactate Dehydrogenase (LDH) is considered a risk factor for overall survival in participants with metastatic melanoma. LDH is a blood test used as a general indicator of the existence and severity of acute or chronic tissue damage and used to monitor cancers such as metastatic melanoma. The baseline LDH value was considered to be the last central laboratory LDH value before randomization. If the central laboratory data was not available, the last non-missing local laboratory value before randomization was used.
  participants
    <0.8 * Upper Limit of Normal (ULN) | 138 | 139 | 277
    0.8-1.1 * ULN | 72 | 69 | 141
    >1.1-2 * ULN | 51 | 56 | 107
    >2 * ULN | 3 | 1 | 4
Metastatic Stage [Number; unit: participants] — Distant Metastatic (M) Stages: MX: Distant metastasis cannot be assessed; M0: No distant metastasis; M1= Distant metastasis; M1a: Metastasis to skin, subcutaneous tissues or distant lymph nodes; M1b: metastasis to lung; M1c: metastasis to all other visceral sites or distant metastasis at any site associated with an elevated serum lactic dehyrogenase
  participants
    M1a | 27 | 21 | 48
    M1b | 66 | 69 | 135
    M1c | 171 | 175 | 346
BRAF Status [Number; unit: participants] — BRAF is a mutation biomarker for melanoma, a human gene that makes the protein B-Raf. The gene is referred to as a protoco-oncogene B Raf and vRaf murine sarcoma viral oncogene homolog B1, while the protein is known as serine/threonine-protein kinase B-Raf. The protein is involved in sending signals inside cells and in directing cell growth. These BRAF mutations were associated with features of high risk melanoma, including truncal primary, earlier age of onset, lack of chronic skin damage and shortened survival. The BRAF statuses included: Wild type and V600E mutation.
  participants
    V 600 E | 65 | 67 | 132
    Wild Type (mutation negative) | 116 | 108 | 224
    unknown | 83 | 90 | 173

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on a Blinded Radiology Assessment of Response Using Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines
Description: PFS was defined as the time from the randomization date to the start of disease progression or patient death, whichever occurred first. Participants who did not have disease progression or had not died were censored at the last known time that the patient was progression free. In the event of palliative radiotherapy or surgery, they were censored at the last assessment where they were documented to be progression-free prior to the date of radiotherapy or surgery. In follow up, participants who began new anticancer therapy prior to documented progression were censored at the last assessment where they were documented as progression free. Those with two or more missing response assessments prior to a visit with documented disease progression (or death) were censored at the last visit where they were documented to be progression free. RECIST defines progressive disease as a ≥ 20% increase taking as reference the smallest sum of the longest diameters recorded since the treatment began.
Time Frame: Response assessment completed every 8 weeks until disease progression for up to 106 weeks; data cut off 30 June 2012
Population: Intent to treat population = The ITT population consisted of all randomized participants regardless of whether the participant received any study drug or had any efficacy assessments collected.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ABI-007 150mg/m^2: ABI-007 150mg/m^2 intravenously over approximately 30 minutes on Days 1, 8 and 15 every 4 weeks
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 264 | 265
months | 4.8 [3.7 to 5.5] | 2.5 [2.0 to 3.6]
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; Two hundred fifty-seven (257) patients were to be randomized to each treatment group for a total of 514 patients. This sample size was chosen to provide at least 80% power for the final analysis (with a two-sided type I error of 0.049) to reject the null hypothesis that the ABI 007/dacarbazine hazard ratio (HR) for PFS is equal to 1.0. This sample size calculation was based on estimates of HR = 0.750. Proportional hazards were assumed; Test type: Superiority or Other; p = 0.044, Log Rank — An interim safety review was performed by DMC. An alpha spending function was utilized to preserve the overall Type 1 error at 0.050. The spending function allocated alpha of 0.001 and 0.049 to the interim and final analyses of PFS, respectively; The treatment difference was tested using the stratified log-rank test, stratified by metastatic stage, region, and baseline LDH; Hazard Ratio (HR) = 0.792, 95.1% CI 2-sided [0.631 to 0.992]

2. Secondary Outcome: Participant Survival
Description: Survival was defined as the time from the date of randomization to the date of death (any cause). Participants were censored at the last known time that they were alive.
Time Frame: Up to 38 months; Up to data cut off of 30 June 2012
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 264 | 265
months | 12.8 [11.3 to 14.6] | 10.7 [9.6 to 12.5]
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; For the participant survival, at the time at least 417 events are recorded, this sample size provides at least 80% power with a two-sided Type 1 error of 0.049 to reject the null hypothesis that the ABI-007/dacarbazine hazard ratio is equal to 1.0. This was based on a HR = 0.760. Proportional hazards were assumed; Test type: Superiority or Other; p = 0.094, Log Rank — At the time of the final PFS analysis, an interim analysis of survival was reported. The spending function allocated an alpha of 0.001 and 0.049 for the interim and final analysis, respectively, to preserve the overall Type I error at 0.050; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.831, 99.9% CI 2-sided [0.578 to 1.196]

3. Other Pre Specified Outcome: Progression-free Survival (PFS) Based on Investigator Assessment Using RECIST Response Guidelines
Description: PFS was defined as the time from the randomization date to the start of disease progression or patient death, whichever occurred first. Participants who did not have disease progression or had not died were censored at the last known time that the patient was progression free. In the event of palliative radiotherapy or surgery, they were censored at the last assessment where they were documented to be progression-free prior to the date of radiotherapy or surgery. In follow up, patients who began new anticancer therapy prior to documented progression were censored at the last assessment where they were documented as progression free. Those with two or more missing response assessments prior to a visit with documented disease progression (or death) were censored at the last visit where they were documented to be progression free.
Time Frame: Response assessments completed every 8 weeks until disease progression; up to data cut off 30 June 2012; 38 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 264 | 265
months | 3.7 [3.1 to 3.9] | 2.1 [1.9 to 2.5]
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; Test type: Superiority or Other; p = 0.086, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.845, 95% CI 2-sided [0.696 to 1.025]

4. Other Pre Specified Outcome: Percent of Participants Who Achieve an Objective Confirmed Complete or Partial Response Based on Blinded Radiology Assessment of Response by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0
Description: RECIST defines complete response (CR): The disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation. All sites must be assessed, including non-measurable sites, such as effusions, or markers. Disappearance of all non-target lesions. The normalization of tumor marker level confirmed at least 4 weeks after initial documentation. Partial response (PR): At least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing. As well as persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Time Frame: every 8 weeks; up to data cut off 30 June 2012
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 264 | 265
percentage of participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 15 | 11
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; Test type: Superiority or Other; p = 0.239, Chi-squared; Response Rate Ratio = 1.305, 95% CI 2-sided [0.837 to 2.035]

5. Other Pre Specified Outcome: Percent of Participants With Stable Disease (SD) for ≥ 16 Weeks, or Confirmed Complete or Partial Response (i.e., Disease Control) Based on a Blinded Radiology Assessment of Response
Description: Disease control is stable disease (SD) for >=16 weeks + complete response (CR) + partial response (PR). See Outcome #4 for definitions of CR and PR.
  RECIST defines SD for target lesions as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: Response assessment completed every 8 weeks until disease progression; up to data cut-off 30 June 2012
Population: ITT
Measure: Number; unit: percent of participants
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 264 | 265
percent of participants | 39 | 27
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; Test type: Superiority or Other; p = 0.004, Chi-squared; Response Rate Ratio = 1.442, 95% CI 2-sided [1.123 to 1.582]

6. Other Pre Specified Outcome: Duration of Response (DOR) in Responding Participants
Description: Duration of response (DOR) as measured by PFS based on radiological review for participants who achieved an objective confirmed response of CR or PR. DOR was defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or participants death from any cause, whichever occurred first. Participants that did not have progression or had not died were censored at the last known time the participant was progression free. Participants that had initiated other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated. Complete response (CR) and partial response (PR) are defined in outcome #4. Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: up to data cut off 30 June 2012
Population: ITT of participants with a confirmed complete or partial overall response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 39 | 30
months | 11.1 [7.3 to NA] — NA = not estimable (ie., the upper bound of survival curve lies above 0.5) | 16.4 [11.0 to 21.8]
Statistical Analysis 1: Comparison: ABI-007 150mg/m^2 vs Dacarbazine 1000mg/m^2; Test type: Superiority or Other; p = 0.057, Log Rank; Hazard Ratio (HR) = 2.201, 95% CI 2-sided [0.959 to 5.053]

7. Secondary Outcome: Summary of Treatment-emergent Adverse Events (AEs)
Description: A Treatment Emergent AE (TEAE) was any AE that began or worsened after the start of the study drug through 30 days after the last dose of study drug or end of study whichever is later. A treatment related toxicity was one considered by the investigator to be possibly, probably or definitely related to study drug. AE's were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V 3.0 criteria and the following scale:
  Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life threatening, and Grade 5 = Death A SAE is any untoward medical occurrence at any dose that is fatal or life threatening, results in persistent or significant disability or incapacity; requires prolonged hospitalizations; is a congenital anomaly birth defect in the offspring of a patient, and conditions not included in the above that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Maximum exposure to study drug was 106 weeks; up to data cut off of 30 June 2012
Population: Treated Population = The Treated population consisted of all randomized participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 257 | 258
participants
  ≥1 TEAE | 255 | 239
  ≥1 TEAE related to study drug | 250 | 212
  ≥1 NCI CTCAE Grade (GR) 3 or above | 167 | 117
  ≥1 NCI CTCAE GR 3 or above TEAE to study drug | 129 | 71
  ≥1 TEAE with outcome of death | 8 | 1
  ≥1 drug related TEAE with outcome of death | 2 | 1
  ≥1 serious TEAE | 62 | 54
  ≥1 serious TEAE related to study drug | 23 | 17
  ≥1 TEAE leading to a dose reduction of study drug | 81 | 51
  ≥1 related TEAE leading to dose reduction | 80 | 49
  ≥1 TEAE leading to drug interruption | 4 | 16
  ≥1 drug related TEAE leading to drug interruption | 3 | 15
  ≥1 TEAE leading to dose delay of study drug | 124 | 84
  ≥1 drug related TEAE leading to dose delay | 106 | 77
  ≥1 TEAE leading to drug discontinuation | 59 | 12
  ≥1 drug related TEAE leading to drug discontinuing | 56 | 11

8. Secondary Outcome: Number of Participants Experiencing Dose Reductions, or Dose Interruptions, or Dose Delays of Study Drug
Description: The number of participants with dose reductions, dose interruptions and dose delays that occurred during the treatment period. Dose reductions, interruptions and delays are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
Time Frame: Maximum study drug exposure 106 weeks; data cut off 30 June 2012
Population: Treated population
Measure: Number; unit: participants
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 257 | 258
participants
  Dose Reductions | 81 | 51
  Dose Interruptions | 6 | 17
  Dose Delay | 145 | 105

9. Secondary Outcome: Nadir for the Absolute Neutrophil Count (ANC) Measurements
Description: Maximal degree of myelosuppression during study drug dosing was represented by the nadir in ANC measurements over all treatment cycles.
Time Frame: Day 1 up to 106 weeks; up to data cut off 30 June 2012
Population: Treated Population = consisted of all randomized participants who received at least one dose of study drug and with at least one post-baseline central laboratory result were included
Measure: Median (Full Range); unit: 10^9/L
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 253 | 246
10^9/L | 1.50 (1.591) [0.1 to 20.0] | 2.40 (1.694) [0.0 to 13.2]

10. Secondary Outcome: Nadir for White Blood Cells (WBCs) Measurements
Description: Maximal degree of myelosuppression was represented by the nadir in white blood cells (WBCs) count measurements over all treatment cycles.
Time Frame: Day 1 up to 106 weeks; up to data cut off 30 June 2012
Population: as for outcome 9
Measure: Median (Full Range); unit: 10^9/L
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 253 | 246
10^9/L | 3.00 (1.934) [0.6 to 22.8] | 4.10 (1.968) [0.5 to 14.7]

11. Secondary Outcome: Nadir for Platelet Count Measurements.
Description: Maximal degree of myelosuppression was represented by the nadir in platelet count measurements over all treatment cycles.
Time Frame: Day 1 up to 106 weeks; up to data cut off 30 June 2012
Population: as for outcome 9
Measure: Median (Full Range); unit: 10^9/L
Groups:
- Dacarbazine Arm B: Dacarbazine 1000mg/m^2 intravenously over approximately 30-60 minutes on Day 1 of each 21 day cycle.
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine Arm B
Number analyzed (Participants) | 252 | 246
10^9/L | 228.5 (71.40) [112 to 437] | 153 (92.01) [9 to 723]

12. Secondary Outcome: Nadir for the Hemoglobin Count Measurements
Description: Maximal degree of myelosuppression during study drug dosing was represented by the nadir in hemoglobin count measurements over all treatment cycles.
Time Frame: Day 1 up to 106 weeks; up to data cut off 30 June 2012
Population: as for outcome 9
Measure: Median (Full Range); unit: g/L
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 253 | 246
g/L | 109.0 [65.0 to 137] | 122.0 [65 to 161]

13. Secondary Outcome: Pharmacokinetic Parameters
Time Frame: On Cycle 1, Day 1 blood samples were taken at 0.25, 3.5, and 24 hr post-infusion end of the initial dose
Population: Patients randomized to receive ABI-007 treatment in Australia, Canada, Europe, United Kingdom and United States had the option to participate in sparse PK sampling in this study. Only 44 participants consented to participate, an insufficient number to support the planned population PK analysis hence these analyses were not performed
Arm/Group | ABI-007 150mg/m^2 | Dacarbazine 1000mg/m^2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Any adverse event (AE) that started at any time from the time the signing of the informed consent to 30 days after the last dose of study drug or End of Study was followed and reported; maximum drug exposure 106 weeks
Groups:
- ABI-007 Arm A: ABI-007 150mg/m^2 intravenously over approximately 30 minutes on Days 1, 8 and 15 of each 28 day cycle
Arm/Group | ABI-007 Arm A | Dacarbazine Arm B
Serious Adverse Events (participants affected / at risk) | 62/257 | 54/258
Other Adverse Events (participants affected / at risk) | 253/257 | 232/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 Arm A (N=257) | Dacarbazine Arm B (N=258)
Pneumonia (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 3 | 4
Erysipelas (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Swine influenza (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Cerebrovascular stenosis (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 5
General physical health deterioration (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Implant site thrombosis (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain 0 1 (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Maculopathy (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 Arm A (N=257) | Dacarbazine Arm B (N=258)
Alopecia (Skin and subcutaneous tissue disorders) | 177 | 9
Rash (Skin and subcutaneous tissue disorders) | 72 | 18
Nail disorder (Skin and subcutaneous tissue disorders) | 52 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 5
Erythema (Skin and subcutaneous tissue disorders) | 16 | 5
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 13
Fatigue (General disorders) | 134 | 110
Oedema peripheral (General disorders) | 54 | 24
Asthenia (General disorders) | 39 | 28
Pyrexia (General disorders) | 32 | 30
Mucosal inflammation (General disorders) | 20 | 13
Pain (General disorders) | 20 | 10
Chills (General disorders) | 12 | 15
Infusion site pain (General disorders) | 2 | 13
Neuropathy peripheral (Nervous system disorders) | 98 | 6
Dysgeusia (Nervous system disorders) | 62 | 24
Peripheral sensory neuropathy (Nervous system disorders) | 52 | 9
Headache (Nervous system disorders) | 42 | 38
Paraesthesia (Nervous system disorders) | 41 | 8
Dizziness (Nervous system disorders) | 32 | 30
Nausea (Gastrointestinal disorders) | 104 | 130
Diarrhoea (Gastrointestinal disorders) | 103 | 45
Constipation (Gastrointestinal disorders) | 83 | 89
Vomiting (Gastrointestinal disorders) | 53 | 56
Abdominal pain (Gastrointestinal disorders) | 34 | 28
Dyspepsia (Gastrointestinal disorders) | 24 | 20
Stomatitis (Gastrointestinal disorders) | 18 | 8
Abdominal pain upper (Gastrointestinal disorders) | 17 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 26
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Upper respiratory tract infection (Infections and infestations) | 18 | 13
Nasopharyngitis (Infections and infestations) | 14 | 10
Neutropenia (Blood and lymphatic system disorders) | 66 | 63
Anaemia (Blood and lymphatic system disorders) | 39 | 28
Leukopenia (Blood and lymphatic system disorders) | 31 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 43
Decreased appetite (Metabolism and nutrition disorders) | 68 | 52
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 10
Insomnia (Psychiatric disorders) | 42 | 31
Anxiety (Psychiatric disorders) | 16 | 19
Weight decreased (Investigations) | 16 | 10
Vision blurred (Eye disorders) | 19 | 6
Lacrimation increased (Eye disorders) | 17 | 4
Flushing (Vascular disorders) | 8 | 16

LIMITATIONS AND CAVEATS:
Participation in the PK sampling for participants randomized to the ABI-007 arm was optional; too few samples were available to support the analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to submission; Celgene shall complete its review within 60 days. Institution shall review comments from Celgene. Upon Celgene's request, proposed publication will be delayed up to 60 additional days to allow Celgene to secure adequate intellectual property protection of patentable material.